CLINICAL TRIAL: NCT04798560
Title: Risk Factors for Pancreaticojejunostomy Leakage Following Whipple Operation
Brief Title: Identifing Risk Factors for Pancreaticojejunostomy Leakage Following Pancreaticoduodenectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dimitrios Vouros (Other)
Responsible Party: Sponsor-Investigator, Dimitrios Vouros, Dr, University of Athens
Organization: University of Athens (Other)
Other Study IDs: 8515/31-05-2019
Record Dates: First submitted 2021-03-02; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Fistula; Whipple Operation; Pancreaticoduodenectomy; POPF
Keywords: pancreaticoduodenectomy; pancreatic cancer; pancreatic adenocarcinoma
MeSH Terms: conditions — Pancreatic Fistula; Pancreatic Neoplasms | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing Whipple operation: After Whipple operation patients will be observed for complications and emphasis will be given on the presence of postoperative pancreatic fistula (POPF) according to the ISGPF 2016 definition. There will be to arms of patients. The first will include patients that do not develop POPF or either develop Biochemical Leak (Grade A). The second group consist of patients that develop either Grade B or Grade C POPF
  Interventions: Procedure: Pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Pancreaticoduodenectomy — Patients udergo pancreaticoduodenectomy for periampullary tumors. All of them are observed for developing POPF

SUMMARY:
Pancreatic cancer is an aggresive type of cancer with poor mean survival rates despite improvements in chemotherapy regimens and advances in surgical techniques. Surgery is the only therapeutic option with an intend to treat. Pancreaticoduodenectomy is indicated for malignancy in the pancreatic head as well as other periampullary tumors. One of the most fatal complications after Whipple operation is postoperative pancreatic fistula as a result of pancreatojejunostomy leakage. Various risk factors for pancreatojejunostomy leakage have been proposed, while there are others less studied.

DETAILED DESCRIPTION:
This is a prospective observational study conducted in the 1st Propaedeutic Department of Surgery of the National and Kapodistrian University of Athens, Greece. Patients with imaging and/or histologically proven periampullary tumors in which Whipple operation is indicated will be enrolled in the study after signing a consent designed by the Hospitals Ethics Commitee and the Department of Surgery. Patients information and medical history will be recorded, giving emphasis on clinical presentation, signs and symptoms related to the patients disease. Laboratory tests will afterwards take place, including biochemical parameters such as total bilirubin levels, serum albumin, CA 19-9, CEA, HbA1c and ferritine levels prior to operation. During operation, as soon as the specimen has been removed, the horizontal and vertical dimension of the pancreatic cutting surface will be measured with the use of an one use sterile ruler and the area of the cutting surface will then be calculated as well as the ratio of the two dimensions (horizontal/vertical). The diameter of the pancreatic duct will be measured either with the same ruler in case diameter is equal or greater than 3mm or with a use of a plastic stent in case diameter is less than 3mm. Pancreatic texture will also be assesed. Other intraoperative datas will be recorded such as the anastomosis technique, duration of surgery, amount of fluid administration, transfusion with fresh frosen plasma or blood units.Postoperatively, amylase from the drains, white blood cell count, platelet count and serum crp levels will be recorded on the 1st, 3rd and 5th postoperative day in all patients. The definition used for postoperative pancreatic fistula (POPF) is based on the International Study Group of Pancreatic Fistula 2016 definition and patients will be categorised accordingly. There will be two arms of patients. The first arm will include patients with either no POPF or Biochemical Leak (BL) and the second arm patients with Grade B or C POPF.

Any complication in the early postoperative period ,defined as the first 30 days after Whipple operation, will be recorded and categorised according to Clavien Dindo classification, including reoperation, readmissions or prolongation of hospital stay. After discharge, follow up of the patients include the EORTC QLQ-C30 and EORTC QLQ-PAN 26 questionnaires that patients have to fill in one, three, six and twelve months after surgery. Reccurence and survival rates will accordingly be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than or equal to 18 years
2. periampullary pathologies (benign or malignant) with indication for panceaticoduodenectomy
3. Pancreaticojejunal anastomosis performed
4. Curative resection
5. Signed informed consent form -

Exclusion Criteria:

1. Age less than 18 years old
2. One stage total pancreatectomy
3. External wirsungostomy without pancreaticojejunal anastomosis
4. Subtotal pancreatectomy without pancreaticojejunal anastomosis
5. Left pancreatectomies
6. Intraoperatively findings of unresectable tumors
7. Pregnancy
8. Concurrent participation in other study(ies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 18 years of age with imaging findings or histologically proven periampullary tumors requiring pancreaticoduodenectomy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Development of Postoperative pancreatic fistula after pancreaticoduodenectomy | 30 days
  Following pancreaticoduodenectomy, patients are observed for developing POPF according to ISGPF definition

SECONDARY OUTCOMES:
Mortality | 30 days
  Mortality rates expressed in % of the patients
Morbidity | 30 days
  Morbidity rates expressed in % of the patients
Postoperative complications | 30 days
  Complications classified according to Clavien-Dindo Classification taking measures from I up to V
Duration of Hospital stay | 60 days
  Duration of Hospital stay in days
Readmission | 30 days
  Readmission rates expressed in % of the patients
Reoperation | 30 days
  Reoperation rates expressed in % of the patients
Overall survival | 2 years
  Estimation of days from operation until death expressed in days

CONTACTS AND LOCATIONS:
Locations (1):
- 1st Propaedeutic Department of Surgery, Hippokrateion General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309
- [Background] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Background] Cullen JJ, Sarr MG, Ilstrup DM. Pancreatic anastomotic leak after pancreaticoduodenectomy: incidence, significance, and management. Am J Surg. 1994 Oct;168(4):295-8. doi: 10.1016/s0002-9610(05)80151-5. PMID 7524375
- [Background] Denbo JW, Orr WS, Zarzaur BL, Behrman SW. Toward defining grade C pancreatic fistula following pancreaticoduodenectomy: incidence, risk factors, management and outcome. HPB (Oxford). 2012 Sep;14(9):589-93. doi: 10.1111/j.1477-2574.2012.00486.x. Epub 2012 May 28. PMID 22882195
- [Background] Nahm CB, Connor SJ, Samra JS, Mittal A. Postoperative pancreatic fistula: a review of traditional and emerging concepts. Clin Exp Gastroenterol. 2018 Mar 15;11:105-118. doi: 10.2147/CEG.S120217. eCollection 2018. PMID 29588609
- [Background] Ryan DP, Hong TS, Bardeesy N. Pancreatic adenocarcinoma. N Engl J Med. 2014 Sep 11;371(11):1039-49. doi: 10.1056/NEJMra1404198. No abstract available. PMID 25207767